CLINICAL TRIAL: NCT03789864
Title: Comparative Analysis of Biodynamic Imaging Utility in Predicting Response to Gemcitabine Chemotherapy for Human and Canine Mycosis Fungoides
Brief Title: Biodynamic Imaging Utility in Predicting Response to Gemcitabine Chemotherapy in Mycosis Fungoides
Acronym: BDI
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of accrual in a timely fashion
Sponsor: Indiana University (Other)
Collaborators: Purdue University (Other)
Responsible Party: Principal Investigator, Lawrence Mark, Charles W. Lewis Investigator and Assistant Professor of Dermatology , Wishard Dermatology Service Chief, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 1804939675
Record Dates: First submitted 2018-12-08; First posted 2018-12-31 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides
Keywords: Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides; Lymphoma

STUDY DESIGN:
Intervention Model Description: This is a single-arm, single-center, non-randomized feasibility study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Individuals undergoing SOC Gemcitabine Treatment for mycosis fungoides (MF) T-cell lymphoma (Other): Standard of Care (SOC) treatment with gemcitabine in this setting is 1200 mg/m2 as a 30 minute infusion given intravenously on days 1, 8, and 15 of every 28-day treatment cycle. Standard dose reductions are expected in patients experiencing unacceptable toxic effects of treatment. All subjects will undergo standardized staging tests, with tumor stage defined according to established guidelines. For this study, three 6-mm x 4-mm dermal punch biopsies from one or more target lesions will be collected prior to treatment initiation and submitted for Biodynamic imaging (BDI). All patients will be considered off-study after completing cycle 2.
  Interventions: Diagnostic Test: Biodynamic imaging (BDI) of mycosis fungoides

INTERVENTIONS:
Diagnostic Test: Biodynamic imaging (BDI) of mycosis fungoides — Skin punch biopsy samples from cutaneous lesions will be profiled for sensitivity to gemcitabine using ex vivo Biodynamic imaging (BDI). A biodynamic profile, of either phenotypic responder or phenotypic non-responder, will be assigned.

SUMMARY:
This is a single-arm, non-randomized feasibility study designed to find out if the laser light-based imaging test called Biodynamic imaging (BDI) can correctly predict the cutaneous T-cell lymphoma mycosis fungoides (MF) cancer response to chemotherapy treatment. The primary objective is to develop phenotypic profiles of response and non-response to gemcitabine, given at a standard-of-care dose and schedule. A secondary objective is to perform a cross-species analysis of phenotypic responses of human and canine mycosis fungoides to gemcitabine using biodynamic imaging. The study will seek to enroll 10 patients with MF who are planning to receive treatment with gemcitabine given at a standard-of-care (SOC) dose and schedule at Indiana University Simon Cancer Center (IUSCC). All subjects will undergo standardized staging tests, with tumor stage defined according to established guidelines. For the study, three 6-mm x 4-mm dermal punch biopsies from one or more target lesions will be collected prior to treatment initiation and sent to Purdue University researchers for BDI. Objective response for tumor samples treated with gemcitabine in the laboratory will be assessed. Patients with an objective response of complete response (CR) or partial response (PR) that persists during the first 2 treatment cycles will be considered to have responsive cancers, while those failing to meet these criteria will be considered to have resistant cancers. All patients will be considered off-study after completing cycle 2. Accrual is expected to last approximately 24 months.

DETAILED DESCRIPTION:
The purpose of this study is to find out if the laser light-based imaging test called Biodynamic imaging (BDI) can correctly predict the response of cutaneous T-cell lymphoma mycosis fungoides cancer to gemcitabine chemotherapy treatment. No untested medications or devices will be used in this study. Subject's response to chemotherapy will be measured after the first and second months (cycles) of chemotherapy; therefore, the BDI test cannot be used to predict whether subject will respond to the treatment or not in advance, and treatment decisions will not be made using any of the information obtained through this study.

As part of routine treatment for mycosis fungoides, subjects who are being referred for routine treatment with gemcitabine chemotherapy given at a standard-of-care (SOC) dose and schedule at the Indiana University Simon Cancer Center (IUSCC) will be enrolled. Standard-of-care Gemcitabine is given intravenously (i.e. in the vein as in infusion) 3 times every 28 days on days 1, 8, and 15. Each 28 day period is called a cycle. Gemcitabine infusion generally lasts 30 minutes. If subject agrees to participate in this study, researchers would document representative skin lesions by color photography including a ruler to estimate the size of the lesion, and objectively calculate disease burden by using the modified Severity Weighted Assessment Tool (mSWAT). Researchers would also collect samples of your tumor tissue before subject starts chemotherapy to be used for the BDI testing in the laboratory by the Purdue University collaborative research team. The BDI testing will be done at baseline on day of collection. We would also evaluate subject's response to treatment after the 1st and 2nd cycles completion through PET/CT or CT scans, skin examinations, and/or laboratory tests depending upon subject's disease. The following is a list of what subjects can expect at each of their study visits.

Pre-treatment: Screening

1. Subject Consenting - approximately 30 - 40 minutes
2. Collect Demographic information, Medical History - approximately 5- 10 minutes
3. Physical Exam/performance status: A physical exam will be performed by the doctor, and the doctor will document subjects' overall health and how well subjects are able to perform their activities of daily living.
4. Skin biopsy: One or more areas of subject's skin that has the cancer will be cleansed with alcohol. The areas will be numbed by injecting a small amount of anesthesia in the skin. As part of routine biopsy procedures in the Department of Dermatology, photographs may be taken of the lesions/tumors that will be biopsied. When the areas of the skin are numb, 3 samples of your skin about 4-mm deep (6-mm wide skin punch biopsies), will be removed from one or more sites and sent for BDI testing. A small stitch will be placed in each biopsy site. Subjects will be given sterile wound dressings and wound care instructions including samples of petrolatum to allow subject to take care of the small wounds. The stitches from the biopsy sites will be removed 10-14 days later.
5. Skin disease severity scoring: In order to determine the extent of subject's disease, the physician will physically examine subject's skin.

Post-Enrollment

1. Laboratory tests: These tests are used to determine subject's fitness to undergo treatment with gemcitabine and to determine extent of disease. These tests are comprehensive metabolic panel (CMP), complete blood count (CBC), and peripheral blood flow cytometry.
2. Scans: Positron emission tomography (PET)/computed tomography (CT) or CT scans of subject's neck, chest, abdomen and pelvis will be done to determine extent of your disease. A PET/CT scan from subject's skull to the base of subject's thighs may be done depending upon subject's disease at the recommendation of subject's doctor.

All of these tests are done routinely in patients with the same disease being referred for treatment with gemcitabine with the exception of skin biopsy and, if needed, flow cytometry and radiological scans after the first round of chemotherapy, which are being done for research purposes. Treatment End of Cycle 1/Before Cycle 2 (Approximately day 28 depending upon whether subjects have any delays in treatment)

1. Physical exam: A routine physical exam will be performed by the doctor.
2. Skin disease severity scoring: The physician will physically examine subject's skin to determine subject's response to chemotherapy at this time point.
3. Laboratory tests: Comprehensive metabolic panel (CMP) and complete blood count (CBC) blood tests will be done as is routine for patients undergoing gemcitabine treatment; however, peripheral blood flow cytometry may also be done depending upon the researcher's assessment of subject's disease to determine subject's response to chemotherapy at this time point.
4. CT scan: A CT scan may also be done depending upon the researcher's assessment of subject's disease to determine subject's response to chemotherapy at this time point.

End of Cycle 2/Before Cycle 3 (Approximately day 56 depending upon whether subject have any delays in treatment)

1. Physical exam: A routine physical exam will be performed by the doctor.
2. Skin disease severity scoring: The physician will physically examine subject's skin to determine subject's response to chemotherapy at this time point.
3. Laboratory tests: Comprehensive metabolic panel (CMP) and complete blood count (CBC) blood tests will be done as is routine for patients undergoing gemcitabine treatment; however, peripheral blood flow cytometry may also be done depending upon the researcher's assessment of subject's disease to determine subject's response to chemotherapy at this time point.
4. CT scan: A CT scan may also be done depending upon the researcher's assessment of subject's disease to determine subject's response to chemotherapy at this time point.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to provide written informed consent and HIPAA authorization
2. Male and female subjects ≥ 18 years of age at the time of informed consent
3. Histologically confirmed diagnosis of mycosis fungoides (MF) T-cell lymphoma
4. Advanced disease as defined by Stage IB (is when ten percent or more of the skin surface is covered with patches, papules, and/or plaques), II-A, II-B, III and IV; disease unresponsive to or contraindicated for skin directed therapy (light treatment, electron beam radiation, topical nitrogen mustards, topical steroids); or otherwise a candidate for systemic therapy due to disease progression
5. Eastern Cooperative Oncology Group (ECOG) performance status score of 0-1
6. Post resolution of all clinically significant toxic effects of prior cancer therapy to Grade ≤ 1 by the National Cancer Institute Common Terminology Criteria for Adverse Events, version 4.03 (NCI-CTCAE, v.4.03)
7. Adequate hematologic and metabolic functions to tolerate gemcitabine.

Exclusion Criteria:

1. Lack of enough skin disease burden to adequately obtain 3 6-mm skin biopsies for ex vivo BDI assessment.
2. Clinical evidence of central nervous system (CNS) metastasis.
3. Psychiatric illness, disability or social situation that would compromise the subject's safety or ability to provide consent, or limit compliance with study requirements
4. Inability or refusal to receive systemic therapy with gemcitabine
5. Prior treatment with gemcitabine
6. Pre-existing allergy to or otherwise contraindicated to receive gemcitabine
7. Patients not on a stable dose of systemic corticosteroid for at least 4 weeks prior to study entry or ≥ 20 mg prednisone daily equivalent
8. Subjects actively on other systemic therapeutic agents for cancer including MF, or would reasonably be expected to receive such treatments during the study period, including ≥ 20 mg prednisone equivalent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2019-10-07 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Development of phenotypic human MF biodynamic profiles | Biopsy samples are collected and imaged prior to each subject's initiation of standard of care gemcitabine treatment
  Dermal punch biopsy samples from subjects' cutaneous mycosis fungoides lesions will be analyzed using ex vivo BDI for sensitivity to gemcitabine. BDI measures intracellular motion patterns (biodynamic profiles) before and after gemcitabine is applied to the sample. Biodynamic profiles associated with poor intercellular organelle motility will be classified as phenotypic responders while those associated with normal intercellular organelle motility will be classified as phenotypic non-responders.

SECONDARY OUTCOMES:
Percent of individual biodynamic profiles with cellular response correlating with individual clinical response. | After day 56 of study for each individual participant
  Correlation against discrete patient outcome classifications (response vs. non-response) will be made to individual biodynamic profiles associated with cellular response vs. non-response.

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence A Mark, MD, PhD, Principal Investigator — Indiana University
Locations (1):
- Indiana University School of Medicine, Department of Dermatology, Indianapolis, Indiana, United States